CLINICAL TRIAL: NCT04491526
Title: Randomized, Quadruple Blinded, Placebo Controlled, Multi-centered Trial Investigating Prophylactic Tamsulosin in Prevention of Postoperative Urinary Retention in Men After Endoscopic Total Extraperitoneal Inguinal Hernia Repair
Brief Title: Study to Prevent Postoperative Urinary Retention
Acronym: STOP-POUR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antonio Nocito, MD (Other)
Responsible Party: Sponsor-Investigator, Antonio Nocito, MD, Professor Antonio Nocito, Director of the Department of General, Visceral and Vascular Surgery and Chief Physician Surgery, Kantonsspital Baden
Organization: Kantonsspital Baden (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-00569
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Urinary Retention; Inguinal Hernia
Keywords: Urinary Retention; Inguinal Hernia Repair; alpha-1 adrenergic receptor antagonists; IPSS
MeSH Terms: conditions — Urinary Retention; Hernia, Inguinal | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin Arm (Experimental): p.o.
  Interventions: Drug: TAMSULOSIN Mepha Ret Depocaps 0.4 mg
- Placebo Arm (Placebo Comparator): p.o.
  Interventions: Drug: Control Intervention

INTERVENTIONS:
Drug: TAMSULOSIN Mepha Ret Depocaps 0.4 mg — 0.4mg/day Tamsulosin hydrochloride ("TAMSULOSIN Mepha Ret Depocaps 0.4 mg") from 5 days prior to the day of surgery, at the day of surgery and for 1 day following surgery. (5+1+1)
  Other Names: Verum
  Arms: Tamsulosin Arm
Drug: Control Intervention — One placebo capsule matching the active study drug per day from 5 days prior to the day of surgery, at the day of surgery and for 1 day following surgery. (5+1+1)
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
Post-operative urinary retention (POUR) is a common complication after inguinal hernia repair with a reported incidence up 34%. It can be described as the inability to initiate urination or properly empty one's bladder following surgery. It is usually self-limited, but it requires the use of catheterization to empty the bladder in order to prevent further injury to the bladder or kidneys and to relief the discomfort of a full bladder. Tamsulosin is a medication that is commonly used in men with urinary symptoms related to an enlarged prostate. There is some evidence to suggest that it may also potentially be beneficial for preventing post-operative urinary retention.

The purpose of this study is to determine if tamsulosin ("TAMSULOSIN Mepha Ret Depocaps 0.4 mg") is effective in preventing post-operative urinary retention following endoscopic total extraperitoneal inguinal hernia repair and its impact on hospital length of stay.

DETAILED DESCRIPTION:
In this RCT subjects are randomly and parallel assigned to one of two groups: one (the experimental group) receiving "Tamsulosin 0.4 mg"/ day, 5 days prior to the day of laparoscopic inguinal hernia repair surgery, at the day of surgery and for 1 day following surgery. (5+1+1), and the other (the control group) receiving one placebo capsule matching the active study drug per day from 5 days prior to the day of surgery, at the day of surgery and for 1 day following surgery. (5+1+1). There will be effective (concealed) randomization of the subjects to the intervention/control groups (to eliminate selection bias and minimize confounding variables). Both groups will be treated identically in all respects except for the intervention being tested and to this end patients, investigators, care providers and outcomes assessors will be blinded to which group an individual is assigned. Group assignment will be performed using a covariate-adaptive allocation procedure to provide a balance for selected covariates (Site, IPSS-Score, Age, "uni- or bilateral surgery" and "history of prostate or bladder surgery". To achieve that; Minimization, first described by Taves [and expanded by Pocock and Simon [the most commonly used covariate-adaptive randomization method will be applied. It achieves the balance in treatment assignments across factor levels by choosing the allocation for the new subject that would lead to the smallest degree of imbalance possible across the set of his baseline characteristics. The two groups are then followed up to 3 days after surgery to see if there are any differences between them in primary and secondary outcomes. Patients are analyzed within the group to which they were allocated, irrespective of whether they experienced the intended intervention (intention to treat analysis). This RCT is designed as a superiority trial and aims to demonstrate the superiority of Tamsulosin in prevention of POUR compared to placebo. We anticipate the detection of a 65% relative risk reduction of POUR in the experimental group in comparison with the placebo group. To detect a 65% reduction of POUR in the experimental group (2.9% anticipated) in comparison with the placebo group (8.3% anticipated) and to assure a study power of 80% with a Fisher's Exact Test and a significance level of 5% and adjusting for a drop-out rate of 2% we need 634 patients in total; 317 in each group. Our target population consists of male patients ≥ 60 yrs, scheduled for elective endoscopic inguinal hernia repair. The studied sample is appropriate to the hypothesis being tested so that any results will be appropriately generalizable.

ELIGIBILITY:
Inclusion Criteria:

* Males
* ≥60 years old
* Planned uni- or bilateral endoscopic total extraperitoneal inguinal hernia repair
* Surgery scheduled more than 6 days from the time of consent
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Orthostatic hypotension (feeling of dizziness after getting up from a sitting or lying position)
* Severe liver disease (Child Pugh C)
* Taking strong inhibitors of CYP3A4 (ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir/ritonavir, lopinavir, or conivaptan)
* Being on alpha-blockers (alfuzosin, doxazosin, prazosin, terazosin, tamsulosin, phenoxybenzamine, or silodosin) or a combination product containing alpha-blocker (duodart)
* History of allergy or sensitivity to tamsulosin or other alpha-blockers (alfuzosin, doxazosin, prazosin, terazosin, or phenoxybenzamine)
* Long term Indwelling urinary or suprapubic catheter
* Status post cystectomy
* Inability to provide informed consent
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Post operative urinary retention (Need for any catheterization postoperatively) | up to 3 days after surgery
  Need for any catheterization postoperatively (Yes/No)

SECONDARY OUTCOMES:
Time to first voiding after surgery | up to 3 days after surgery
  secondary outcomes in Non-POUR Patients
Urinary Volume measurement at defined points in time (n) | up to 12 hours after surgery
  secondary outcomes in all Patients
Volume of first micturition after surgery | up to 12 hours after surgery
  secondary outcomes in Non-POUR Patients
Post-operative Pain (Quantity of Pain / VAS-Score) | up to 3 days after surgery
  Quantity of pain is verified at arrival in the PACU and at every 6 hours by the nursing staff, using the standardised numeric rating scale. The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older.
Need for opioid analgesics post operatively | up to 3 days after surgery
  secondary outcomes in all Patients
Quantity of post-operative opioid use (opioid dosage will be converted to oral morphine equivalence dose) | up to 3 days after surgery
  opioid use is documented in the patient's record, opioid dosage will be converted to oral morphine equivalence dose
Intraoperative applications of opioid analgesics (Yes/No) | intra-operative period
  Opioid use during surgery is documented in the patient's record, this is a binary endpoint opioid use; (yes/ no)
Quantity of intra-operative opioid use opioid dosage will be converted to oral morphine equivalence dose) | intra-operative period
  Opioid use during surgery is documented in the patient's record, opioid dosage will be converted to oral morphine equivalence dose
Amount of intraoperative fluid administration | intra-operative period
  Intraoperative fluid administration (in milliliter) is documented in the patient's record
International Prostate Symptom Score (IPSS score) pre-surgery (-5d) | min. 5 days prior to surgery
  0-7 Mildly symptomatic / 8-19 Moderately symptomatic / 20-35 Severely symptomatic
International Prostate Symptom Score (IPSS score) post-surgery (3d) | 3 days post surgery
  0-7 Mildly symptomatic / 8-19 Moderately symptomatic / 20-35 Severely symptomatic
Change in International Prostate Symptom Score (IPSS score) from baseline prior to surgery (-5d) to day 3(+3d) after surgery | 3 days post surgery
  0-7 Mildly symptomatic / 8-19 Moderately symptomatic / 20-35 Severely symptomatic
Side-effects of study medication (orthostatic hypotension, retrograde ejaculation, Floppy-Iris-Syndrom) | 5 days prior to surgery (-5d) to day 3(+3d) after surgery
  Will be documented in the patient record by the study personnel, binary endpoint (Yes/No)
In hospital complications (using the evaluated standard classification for complication in surgery (Classification Grade I-V) ) | as long as the patient is labeled inpatient, on average 1-3 days
  secondary outcomes in all Patients
Length of hospital stay in days (Inpatients) | as long as the patient is labeled inpatient, on average 1-3 days
  secondary outcomes in all Patients
Time to discharge after surgery in hours (outpatients) | up to 12 hours after surgery
  secondary outcomes in all Patients
Residual urinary volume after catherization | up to 12 hours after surgery
  secondary outcomes in POUR Patients
Macrohematuria | 3 days post surgery
  secondary outcomes in POUR Patients
Relevant injury to the urethra (Presence of a Via falsa diagnosed by a urologist) | 3 days post surgery
  secondary outcomes in POUR Patients
Catheter-related infections | 3 days post surgery
  secondary outcomes in POUR Patients
Catheter-related bladder discomfort ( (Ggrading according to the 3three Ggrades (mild, moderate, severe) | 3 days post surgery
  secondary outcomes in POUR Patients
Prostatitis | 3 days post surgery
  secondary outcomes in POUR Patients
Failed first trial without catheter (TWOC: need for a second catheter insertion due to insufficient voiding after TWOC). | 1 day post surgery
  secondary outcomes in POUR Patients

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Nocito, Prof, Principal Investigator — Kantonsspital Baden AG, Im Ergel 1, 5404 Baden, Switzerland
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data are available upon reasonable request from https://orcid.org/0000-0002-7339-1458.

REFERENCES:
- [Derived] Bieri U, Slieker J, Hefermehl LJ, Soppe S, Teufelberger G, Tedaldi R, Graf N, Bieri M, Nocito A. Randomised, quadruple blinded, placebo controlled, multicentre trial investigating prophylactic tamsulosin in prevention of postoperative urinary retention in men after endoscopic total extraperitoneal inguinal hernia repair (STOP-POUR trial): a study protocol. BMJ Open. 2021 Dec 7;11(12):e048911. doi: 10.1136/bmjopen-2021-048911. PMID 34876420